CLINICAL TRIAL: NCT06411951
Title: Integrated Care After Repeated Psychiatric Hospital Stays (INTUK) - Evaluation of an Interdisciplinary Treatment Program
Brief Title: Integrated Care After Repeated Psychiatric Hospital Stays - Evaluation of an Interdisciplinary Treatment Program
Acronym: INTUK
Status: Enrolling by invitation | Type: Observational
Sponsor: Michael Rufer (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Michael Rufer, Prof. Dr. med. Michael Rufer, Triaplus AG Klinik Zugersee - Zentrum für Psychiatrie und Psychotherapie
Organization: Triaplus AG Klinik Zugersee - Zentrum für Psychiatrie und Psychotherapie (Other)
Other Study IDs: 2023-00836
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: High Utilization / Heavy Use; Psychiatric Hospitalization; Rehospitalization; Intensive Care Psychiatric Disorder; Chronic Psychiatric Disorder; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Participation in the INTUK care offer at Klinik Zugersee — Person-centered treatment and care tailored to the individual patients needs by a team consisting of a senior physician, a nurse, social workers and peers.

SUMMARY:
The study aims to evaluate the treatment effects as well as inhibiting and promoting factors in the implementation of the new INTUK care offer in a sample of "heavy users", i.e. psychiatric patients with 4 or more prior inpatient admissions at Klinik Zugersee, by means of a longitudinal, prospective-retrospective study. For this purpose, medical records will be analysed and participants will be asked to fill out questionnaires addressing different aspects of mental health, quality of life and patient satisfaction. In addition, semi-structured interviews will be conducted with a subset of patients as well as staff members of the INTUK care offer.

DETAILED DESCRIPTION:
In the mental health literature, the terms "heavy users" or "high utilizers" have been coined to describe a relatively small group of people with chronic mental illness, with excess use of inpatient psychiatric services. Although these terms are used both nationally and internationally, there is no consensus on how they are defined. For example, in Switzerland, they are used by the Swiss Health Observatory (Obsan) and the Federal Office of Public Health. Previous research suggests that even though only 10% to 30% of all inpatients qualify as "heavy users", their use of the healthcare system's resources is well above average. In German-speaking countries, there are currently only a few scientific studies on this group of patients, especially on the question of which offers are best suited to better integrate existing models of care, and how to make them more effective. Due to the separate enumeration of outpatient and inpatient care in Switzerland (as in many other countries), integrated models of care that are particularly needed for this group of patients are currently lacking. This can result in costly under- and incorrect treatment with more frequent discontinuations. In addition, apart from the treatment of medical issues, other aspects often play an important role in the care of chronically ill patients, such as socio-economic difficulties (e.g. in the areas of work and housing or financial problems). Therefore, in the recently completed National Research Program (NRP) 74 "Healthcare" of the Swiss National Science Foundation, the numerous interfaces between care settings were identified as a central field of action, which is a particularly the case in patients with chronic illnesses: "In the highly specialized, decentralized health care system in Switzerland, coordination between multiple medical and non-medical services is difficult."

INTUK (Integrated care after repeated psychiatric hospital stays) represents a new interprofessional and integrated care program at Klinik Zugersee, which aims to bridge such interfaces and improve the treatment of people with chronically recurrent mental illness. A team consisting of a senior physician, nurse, social worker, and peer will deliver person-centered care tailored to individual needs in these mostly complex care situations. Contact is initiated with the affected patients during their inpatient stay to build relationships and increase motivation for subsequent, individually planned treatment and care. For example, round-table discussions can take place with the specialists and community-based providers involved in the follow-up treatment before the patient is discharged. After discharge, the same team continues to provide support and coordinate access to outpatient and semi-inpatient treatment, counselling and self-help services. In the case of social difficulties, social work coaching or accompaniment to offices and social institutions takes place will be provided. Another service is the joint drafting of a psychiatric living will to determine consent and rejection for future psychiatric treatments. Wherever possible, close others and the wider social environment are also included in consultation with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric patients with 4 or more inpatient admissions at Klinik Zugersee in the past 24 months.

Exclusion Criteria:

* Age < 18 years.
* Lack of written informed consent.
* Incapability of judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients with 4 or more inpatient admissions at Klinik Zugersee in the past 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Admission rate | 01.06.2023 - 31.05.2027
  Participation in the INTUK program will be associated with a significant change in the total number of inpatient admissions.

SECONDARY OUTCOMES:
Length of hospital stays | 01.06.2023 - 31.05.2027
  Participation in the INTUK program will be associated with a change in the total length of hospital stays (measured in days).
Treatment effects | 01.06.2023 - 31.05.2027
  Participation in the INTUK program will be associated with a significant change in the impairment due to psychiatric symptoms measured using the Symptom-Checkliste-K-9 (SCL-9-K; on a numeric scale from 9 to 36; higher indicating a worse outcome).
Treatment effects | 01.06.2023 - 31.05.2027
  Participation in the INTUK program will be associated with a significant change in the quality of life measured using the World Health Organization Quality of Life Brief Version (WHOQOL-BREF; on a numeric scale of 0 to 100, lower indicating a worse outcome).
Treatment effects | 01.06.2023 - 31.05.2027
  Participation in the INTUK program will be associated with a significant change in the severity of the mental illness measured using the Global Clinical Impression Scale (CGI; on a numeric scale from 1 to 7; higher indicating a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rufer, Prof. Dr., Principal Investigator — Triaplus AG - Klinik Zugersee
Locations (1):
- Triaplus AG - Klinik Zugersee, Oberwil, Canton of Zug, Switzerland

IPD SHARING:
Plan to Share IPD: No